CLINICAL TRIAL: NCT03157479
Title: Intraoperative Protective Ventilation for Obese Patients Undergoing Gynaecological Laparoscopic Surgery. A Single-centre Randomized, Controlled Trial
Brief Title: Intraoperative Protective Ventilation for Obese Patients Undergoing Gynaecological Laparoscopic Surgery
Acronym: Inprove4large
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Massimo Antonelli, MD, Full Professor, Director of the Department of Anesthesiology and Intensive Care Medicine, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: InproveForLarge
Record Dates: First submitted 2017-05-12; First posted 2017-05-17 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Anesthesia; Surgery--Complications
Keywords: Mechanical ventilation
MeSH Terms: interventions — Anesthetics, Intravenous; Crystalloid Solutions; Lung Volume Measurements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protective ventilation (Experimental): Volume controlled ventilation with tidal volume 6-7 ml/kg of predicted body weight (45.5 + 0.91 (height [cm] -152.4)), FiO2 0.4 and PEEP 10 cmH2O during the whole study period. Respiratory rate will be titrated to keep end-tidal CO2 values between 30 and 40 mmHg. I:E ratio will be set in order to obtain an inspiratory time of 0.8 seconds and an inspiratory pause of 0.3 seconds and FiO2 will be kept unchanged during the whole study period. In patients in this group, recruiting maneuvers will be performed throughout a stepwise 5 cmH2O PEEP increase every 30 seconds to achieve a PEEP of 35 cmH2O during Pressure Controlled Ventilation (10 cmH2O of inspiratory pressure while keeping respiratory rate unmodified), followed by a stepwise 5 cmH2O PEEP reduction every 30 seconds until the baseline set peep is reached.
  Interventions: Drug: Intravenous anesthetic; Drug: Crystalloid Solutions; Diagnostic Test: Esophageal pressure measurement; Diagnostic Test: Lung volume measurement with the nitrogen washin-washout technique
- Standard Ventilation (Active Comparator): Volume controlled ventilation with tidal volume 10 ml/kg of PBW (45.5 + 0.91 (height [cm] -152.4)), FiO2 0.4 and PEEP 5 cmH2O during the whole study period. Respiratory rate will be titrated to keep end-tidal CO2 values between 30 mmHg and 40 mmHg. I:E ratio will be set in order to obtain an inspiratory time of 0.8-1 seconds and an inspiratory pause of 0.3 second
  Interventions: Drug: Intravenous anesthetic; Drug: Crystalloid Solutions; Diagnostic Test: Esophageal pressure measurement; Diagnostic Test: Lung volume measurement with the nitrogen washin-washout technique

INTERVENTIONS:
Drug: Intravenous anesthetic — Anaesthesia induction will be obtained with i.v. 2-3 mg/kg propofol, 0,6-0,8 mcg/kg fentanyl, and 0.9-1,2 mg/kg rocuronium. Anaesthesia will be maintained with i.v. propofol continuous infusion, with a dose titrated to achieve a bi-spectral index value between 40 and 50
Drug: Crystalloid Solutions — Balanced crystalloids will be administered to patients in both groups as a standard rate of 3-5 ml/kg/h. Treatment of eventual hemodynamic instability will be left to the attending physician
Diagnostic Test: Esophageal pressure measurement — A nasogastric polyfunctional tube (Nutrivent, Sidam, Italy) will be placed after anaesthesia induction in all enrolled patients to measure esophageal pressure, estimate pleural pressure and compute transpulmonary pressure
Diagnostic Test: Lung volume measurement with the nitrogen washin-washout technique — Lung volume will be measured through nitrogen wash-in wash-out technique and low-flow Pressure-volume curve will be recorded to estimate differences in alveolar recruitment between the two study groups.

SUMMARY:
Background. The use of a comprehensive strategy providing low tidal volumes, peep and recruiting maneuvers in patients undergoing open abdominal surgery improves postoperative respiratory function and clinical outcome. It is unknown whether such ventilatory approach may be feasible and/or beneficial in patients undergoing laparoscopy, as pneumoperitoneum and Trendelenburg position may alter lung volumes and chest-wall elastance.

Objective. The investigators designed a randomized, controlled trial to assess the effect of a lung-protective ventilation strategy on postoperative oxygenation in obese patients undergoing laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for gynaecological laparoscopic surgery in the Trendelenburg position
* Obesity with body mass index>35 kg/m^2
* written informed consent

Exclusion Criteria:

* Clinical history or signs of chronic heart failure
* history of neuromuscular disease
* history of thoracic surgery
* pregnancy
* chronic respiratory failure requiring long-term oxygen administration

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Postoperative oxygenation | One hour after extubation
  PaO2/FiO2 ratio 1 hour after extubation, while the patient is receiving oxygen through VenturiMask 40%

SECONDARY OUTCOMES:
Postoperative forced expiratory volume in 1 second (FEV1) | 48 hours after the end of surgery
  volume exhaled during the first second of a forced expiratory maneuver started from the level of total lung capacity
Postoperative forced vital capacity (FVC) | 48 hours after the end of surgery
  the total amount of air exhaled during a forced expiratory maneuver started from the level of total lung capacity
Postoperative Tiffeneau index | 48 hours after the end of surgery
  computed as FEV1/FVC
Postoperative Dyspnea | 1 hour after surgery
  Dyspnea assessed by Borg dyspnea scale
Pulmonary infection | 24 hours after the end of surgery
  modified clinical pulmonary infection score (mCPIS)
Postoperative pulmonary infiltrates | 24 hours after the end of surgery
  Evaluated with the chest x-ray by two independent clinicians blinded to treatment assignment
Intraoperative driving pressure | during surgery, recorded on a 60-minute basis
  driving pressure, computed as Plateau pressure-PEEP
Intraoperative lung driving pressure | during surgery, recorded on a 60-minute basis
  transpulmonary driving pressure, computed as Transpulmonary end-inspiratory pressure-transpulmonary total end-expiratory pressure
Intraoperative oxygenation | during surgery, recorded on a 60-minute basis
  PaO2/FiO2
Intraoperative dead space | during surgery, recorded on a 60-minute basis
  Approximated as the difference between End-tidal CO2 and PaCO2 divided by PaCO2
Lung recruitment | during surgery, recorded on a 60-minute basis
  lung recruitment/changes in end expiratory lung volume between the two groups
Intraoperative blood pressure | during surgery, recorded on a 60-minute basis
  Arterial blood pressure
Intraoperative respiratory system compliance | during surgery, recorded on a 60-minute basis
  computed as Tidal volume/airway driving pressure
Intraoperative lung compliance | during surgery, recorded on a 60-minute basis
  computed as Tidal volume/lung driving pressure

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Antonelli, MD, Principal Investigator — Catholic University of the Sacred Heart
Locations (1):
- General surgery OR, A. Gemelli hospital, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Grieco DL, Russo A, Anzellotti GM, Romano B, Bongiovanni F, Dell'Anna AM, Mauti L, Cascarano L, Gallotta V, Rosa T, Varone F, Menga LS, Polidori L, D'Indinosante M, Cappuccio S, Galletta C, Tortorella L, Costantini B, Gueli Alletti S, Sollazzi L, Scambia G, Antonelli M. Lung-protective ventilation during Trendelenburg pneumoperitoneum surgery: A randomized clinical trial. J Clin Anesth. 2023 May;85:111037. doi: 10.1016/j.jclinane.2022.111037. Epub 2022 Dec 7. PMID 36495775